CLINICAL TRIAL: NCT03681210
Title: Destination Therapy Post Approval Study
Acronym: DT PAS
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: DT PAS
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Heart Failure
Keywords: Heart Failure; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients implanted with HVAD System: Patients intended to be implanted with a HVAD for use as destination therapy are eligible for enrollment into the DT PAS and must be consented for the study prior to the HVAD implant.
  Interventions: Device: HeartWare Ventricular Assist Device

INTERVENTIONS:
Device: HeartWare Ventricular Assist Device — The HVAD is an implantable centrifugal rotary blood pump that is implanted in the pericardial space and is designed to provide up to 10 L/min of blood flow from the left ventricular to the aorta. The HVAD System is comprised of three major components: the HVAD (pump) with inflow and outflow conduits, a Controller (microprocessor unit that controls the operation of the HVAD), and power sources (AC and DC power adapters that provide power to the Controller and implanted HVAD).
  Other Names: HVAD

SUMMARY:
Medtronic is sponsoring the HeartWare™ HVAD™ Destination Therapy (DT) Post Approval Study (PAS) to further confirm safety and effectiveness of the HeartWare Ventricular Assist Device System (HVAD System) when used as intended, in "real-world" clinical practice.

The Destination Therapy Post Approval Study (DT PAS) is conducted within Medtronic's Product Surveillance Platform.

DETAILED DESCRIPTION:
The HeartWare Destination Therapy (DT) Post Approval Study (PAS) is a prospective, observational, multi-site study. Enrollment into the DT PAS will be comprised of newly enrolled, commercial use DT patients with the HeartWare Ventricular Assist Device System (HVAD System). Patients enrolled in DT PAS will be followed for 5 years post-implant or until study closure, patient death, patient exit from the PAS (i.e., withdrawal of consent), or patient has HVAD device removed without replacement (i.e., transplant, recovery) or device is exchanged for non-HVAD. The total estimated study duration is approximately 7 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient is intended to receive or be treated with a HeartWare HVAD System for use as destination therapy
* Patient is consented prior to the HVAD implant procedure

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results (i.e., no required intervention that could affect interpretation of all-around product safety and or effectiveness)
* Patient less than 18 years of age.
* Patient with previous support by long-term mechanical circulatory support (MCS), not including temporary mechanical circulatory support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients intended to be implanted with a HVAD for use as a destination therapy are eligible for enrollment into the DT PAS and must be consented for the PAS prior to the HVAD implant. The PAS cohort will be comprised of 300 newly enrolled PAS patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Long-term complication free survival | Implant to 2 years
  Complications include death, disabling stroke, or device malfunction or failure requiring exchange, explantation or urgent transplantation.

SECONDARY OUTCOMES:
Rate of stroke | Implant to 2 years
  The rate of stroke on device will be analyzed using Kaplan-Meier methods.
Rate of late stroke | 2 years post-implant to 5 years
  The rate of late stroke on device will be analyzed using Kaplan-Meier methods for those surviving stroke-free for 24 months post-implant.
Stroke severity | Occurrence of stroke to 24 weeks post-stroke
  Modified Rankin Scale (mRS) scores will be collected at the time associated with stroke on device and at 12 and 24 weeks post-stroke. The distribution of mRS scores for all strokes occurring in the study will be presented, separating stroke occurring prior to 24 months post-implant and those occurring greater than 24 months post-implant.

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - Saint Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - University of California San Diego, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Stanford University Hospital, Stanford, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Coral Gables, Florida
  - Mayo Clinic (Jacksonville FL), Jacksonville, Florida
  - AdventHealth, Orlando, Florida
  - University of South Florida Health, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Advocate Christ Medical Center (Cardiac Surgery Clinical Research Center), Oak Lawn, Illinois
  - Saint Vincent Medical Group, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Medical Center, New York, New York
  - Columbia University, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - The Lindner Christ Hospital, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - PennState Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute Dallas - Baylor University Medical Center (BUMC), Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Sciences Center, Houston, Texas
  - Methodist Hospital San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No